CLINICAL TRIAL: NCT06710015
Title: B.Fert: Retrospective and Prospective Observational Study on Fertility Parameters in Women With Germline Variants in BRCA1 and BRCA2
Brief Title: Study on Fertility Parameters in Women With Germline Variants in BRCA1 and BRCA2
Acronym: BFert
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Lucci Cordisco Emanuela, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6591
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: BRCA1 and/or BRCA2 Variant Carriers; Fertility; Reproductive Age; Menopause; Pregnancy Outcomes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- BRCA1 and BRCA2 carriers: Inclusion criteria:
  * age > 18 years
  * presence of a pathogenic variant in the BRCA genes
  * signed informed consent for study participation
- Control cohort: * >18 y.o
  * Relatives up to the third degree of kinship from cohort 1 who tested negative on predictive testing for the familial pathogenic variant in the BRCA genes, matched for age where possible.

SUMMARY:
Pathogenic variants (PVs) in the BRCA1 and BRCA2 genes are associated with an increased risk of developing breast and ovarian cancers. According to current guidelines from the National Comprehensive Cancer Network, the risk of developing breast cancer exceeds 60% for both genes, while the risk for ovarian cancer ranges from 39% to 58% for the BRCA1 and from 13% to 29% for the BRCA2. The detection of a pathogenic variant in the BRCA1 or BRCA2 genes necessitates both the establishment of appropriate primary and secondary surveillance measures for carriers and the discussion of the familial implications of such findings.

The molecular basis initially suggesting a possible association between germline variants in BRCA1 and BRCA2 genes and diminished ovarian reserve lies in the cellular impact of impaired or defective repair of DNA double-strand breaks (DSBs) on oocytes. Notably, BRCA1 and BRCA2 genes play a key role in the ATM-related mechanism for DSB repair through the homologous recombination (HR) pathway.

Although preclinical evidence supports a potential correlation between defective DSB repair and normal follicle maturation processes, clinical studies on large cohorts of patients with pathogenic BRCA1 and BRCA2 variants yield inconsistent results. This discrepancy is likely attributable to the inherent challenges in recruiting a sufficiently homogeneous and statistically significant sample size.

The aim of the study is to evaluate reproductive capacity in women carrying pathogenic variants in the BRCA1/2 genes by assessing the number of pregnancies during the period from January 1, 2018, to December 31, 2023. Secondary objectives include evaluating menopausal characteristics and pregnancy outcomes.

ELIGIBILITY:
BRCA1 and BRCA2 carriers

Inclusion Criteria:

* age > 18 years
* presence of a pathogenic variant in the BRCA genes
* signed informed consent Exclusion Criteria
* presence of a pathogenic variant in another gene (not BRCA)
* significant psychiatric or clinical impairment affecting the ability to consent to the study

Control cohort

Inclusion Criteria:

- Relatives up to the third degree of the first cohort who tested negative on predictive testing for the familial pathogenic variant in the BRCA genes, matched for age where possible.

Exclusion Criteria:

* absence of a pathogenic variant in another gene (non-BRCA) found in a family member
* significant psychiatric or clinical impairment affecting the ability to consent to the study

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Carriers and non carriers of BRCA pathogenic variants
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the reproductive capacity in women carrying PVs in BRCA1/2 genes | 1 year
  Evaluate number of pregnancies

SECONDARY OUTCOMES:
The evaluation of menopausal characteristics and pregnancy outcomes | 1 year
  Evaluate: age at menopause, type of menopause, number of miscarriages, age at pregnancies, cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Lucci Cordisco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Genetica Medica Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No